CLINICAL TRIAL: NCT00195806
Title: Divalproex Sodium Extended-Release Tablets for Migraine Prophylaxis in Adolescents: An Open-Label, Long-Term Safety Study
Brief Title: Study Designed to Evaluate the Safety of Prophylactic Depakote ER in the Treatment of Adolescents With Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M03-648
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2007-09-03 (Estimated); Status verified 2007-08

CONDITIONS: Migraine
Keywords: Migraine; Depakote ER; Divalproex sodium
MeSH Terms: conditions — Migraine Disorders | interventions — Valproic Acid

INTERVENTIONS:
Drug: divalproex sodium

SUMMARY:
The purpose of this study is to determine if long-term treatment, up to 1 year, with Depakote ER is safe in the reduction of occurrence of migraine headaches in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Subject and subject's legal representative have voluntarily signed and dated an IRB-approved informed assent form and an IRB-approved informed consent form, respectively, before any study-specific procedures or tests are performed;
* Subject is male, or a non-pregnant, non-lactating female;
* Subject is between 12 and 17 years of age, inclusive, at the Screening Visit;
* Subject weighs at least 77 lbs. (i.e., 35 kg);
* Subject currently has diagnosis of migraine headaches consistent with International Headache Society (IHS) criteria;
* Subject is judged to be in generally good health based on the results of a medical history, physical examination, 12-lead electrocardiogram (ECG), and laboratory profile; and
* In the investigator's opinion, the subject will benefit from Depakote ER for migraine prophylaxis.

Exclusion Criteria:

* History of allergic reaction or significant sensitivity to valproate or similar drugs;
* History of noncompliance with medication or medical instructions;
* Recent (previous 6 months) history of drug and/or alcohol abuse or has a positive urine drug screen, at the Screening Visit, for drugs of abuse (e.g., amphetamines, barbiturates, benzodiazepines, cocaine, opiates, and phencyclidine [PCP]);
* Female, of childbearing potential, and not using an effective method of birth control (e.g., total sexual abstinence or contraceptives) as judged by the investigator.
* Use of the following medication classes or any specific drug listed below:

  * anti-depressants, other antiepileptic drugs (AEDs)
  * aspirin and/or aspirin-containing products
  * chronic use of systemic corticosteroids, clonazepam,diazepam, erythromycin, ethosuximide, pemoline, phenobarbital,rifampin,tolbutamide, zidovudine
  * anticoagulant drug therapy;
* Any serious medical or psychiatric disorder(s), including epilepsy and obesity, that may confound the interpretation of the results from this study;
* Central nervous system (CNS) neoplasm, CNS infection, demyelinating disease, degenerative neurological disease, or any progressive CNS disease;
* History of encephalopathy, hepatitis, pancreatitis, or urea-cycle disorder or any underlying condition/disease, which might interfere with study drug absorption or completion of study drug therapy evaluation throughout the duration of the trial;
* Screening laboratory results indicate the presence of Hepatitis B surface antigen (HBsAg), or Hepatitis C antibody or known history of any positive test result for HIV;
* Screening laboratory results indicate:

  1. Platelet count =/< 100,000/uL
  2. ALT or AST =/> 2 times Upper Limit of Normal (ULN);
* Receipt of an investigational drug within 30 days prior to study drug administration or scheduled to receive any other investigational drug anytime during the study;
* Participation in a prior Depakote ER migraine study (M02-488 or M02-554); or if for any reason, subject is considered by the investigator to be an unsuitable candidate to receive Depakote or to participate in this study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 315
Dates: Start 2005-02

PRIMARY OUTCOMES:
Number of migraine headache days

SECONDARY OUTCOMES:
Adverse events
Laboratory data
Vital signs
Study drug exposure
Behavioral/cognitive assessments

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information 800-633-9110, Study Director — Abbott
Locations (1):
- Global Medical Information - Abbott, North Chicago, Illinois, United States